CLINICAL TRIAL: NCT01073852
Title: Hydroxychloroquine Efficacy in Chronic Urticaria
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn, not funded
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Michael Fahrenholz, MD, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pending
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Urticaria
Keywords: Chronic Urticaria; Hives; Hydroxychloroquine
MeSH Terms: conditions — Chronic Urticaria; Urticaria | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will be taking placebo medication throughout study.
  Interventions: Drug: Placebo
- Hydroxychloroquine (Active Comparator): Patients will be taking hydroxychloroquine throughout study.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Placebo — Placebo pill, 1 pill orally twice daily for 9 weeks.
  Arms: Placebo
Drug: Hydroxychloroquine — Patients will be taking hydroxychloroquine 200mg orally twice/daily.
  Arms: Hydroxychloroquine

SUMMARY:
This study is for those people with difficult to treat hives. We are investigating whether or not a different medication, hydroxychloroquine, works to treat a certain type of hives. Hydrochloroquine is currently approved by the Food and Drug Administration (FDA), for treating arthritis, therefore it is considered investigational in this study.

Hypothesis: Hydroxychloroquine will prove to have an efficacious response in terms of Urticarial Symptoms, on patients with chronic urticaria.

DETAILED DESCRIPTION:
Our research question is: Is hydroxychloroquine an efficacious medicine to use in patients with chronic urticaria? Answering this question should help allergists treat chronic urticaria with a more evidence based approach. To date there has one been one prospective trial evaluating hydroxychloroquine in hives, and although it showed a trend towards efficacy (0.05<p<0.10), it was not statistically significant. There have been case series, and anecdotal reports which seem to demonstrate efficacy of chloroquine in chronic urticaria. Because of these reports hydroxychloroquine is often the first medication used in patients with chronic hives that are refractory to standard therapy of antihistamines. We believe an evidence based answer to this question will be an important step towards improved treatment of this disease.

We plan to ascertain the efficacy of hydroxychloroquine by completing a randomized double blinded placebo controlled study of treatment in patients with chronic urticaria. We will be measuring an Urticarial Score to evaluate hive symptoms. We will be measuring them at baseline, and at the end of the study to note change in drug vs placebo.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion:

  1. Age >18, Age<65
  2. Chronic Urticaria refractory to treatment with standard anti-histamines
  3. Minimum Urticaria Score

Exclusion Criteria:

* Exclusion:

  1. Pregnancy
  2. Vasculitis
  3. Trigger Induced Urticaria
  4. Food intolerance
  5. Malignancy
  6. Kidney or liver dysfunction
  7. Systemic diseases
  8. Hypersensitivity to hydroxychloroquine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Urticarial Symptom Score | 10 weeks

SECONDARY OUTCOMES:
Difference in Basophil Activation | 10 weeks
Difference in Rescue Medication Usage | 10 weeks
Difference in Dermatology Life Quality Index | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pogie Pongonis, MD, Principal Investigator — Vanderbilt University; John Fahrenholz, MD, Study Director — Vanderbilt University

REFERENCES:
- [Background] Reeves GE, Boyle MJ, Bonfield J, Dobson P, Loewenthal M. Impact of hydroxychloroquine therapy on chronic urticaria: chronic autoimmune urticaria study and evaluation. Intern Med J. 2004 Apr;34(4):182-6. doi: 10.1111/j.1444-0903.2004.00532.x. PMID 15086698